CLINICAL TRIAL: NCT07324915
Title: Effect of Buzzy Bee to Reduce Pain Perception During Inferior Alveolar Nerve Block in Children - A Cross Over Study
Brief Title: EFFECT OF BUZZY BEE TO REDUCE PAIN PERECEPTION DURING INFERIOR ALVEOLAR NERVE BLOCK IN CHILDREN - A CROSS OVER STUDY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, satish vishwanathaiah, Associate professor, University of Jazan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COLLEGE OF DENTISTRY jazan
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUZZY BEE (Experimental): Vibrating device
  Interventions: Device: BUZZY BEE [ Vibrating device]
- Conventional technique (Active Comparator): conventional way
  Interventions: Device: Conventional technique

INTERVENTIONS:
Device: BUZZY BEE [ Vibrating device] — already described
  Other Names: EXPERIMENTAL
  Arms: BUZZY BEE
Device: Conventional technique — described
  Arms: Conventional technique

SUMMARY:
Pain management during invasive dental procedures is crucial to avoid noncompliance and treatment avoidance. Thus, measures to reduce injection discomfort are needed to prevent patients from avoiding dental treatment. Tooth extractions, and invasive dental procedures cause pain. Local anesthetics are one of the most effective and safest pain relievers. Even though many children have needle fear, anesthetic may still be uncomfortable. Fear of pain, especially in young children, is real since it affects health outcomes. Anxiety and fear may delay dental treatment and harm the patient's oral health. Distraction, topical anesthetic gel, modifying infiltration rate, intra-oral vibrating devices, computerized delivery systems, pre-cooling injection site, and other pharmacological, physical, and psychological interventions have all been proposed as potential pain relievers. An example of this kind of system One approach that combines an extraoral cold with a vibrating device is Buzzy Bee.

DETAILED DESCRIPTION:
Before start of the study a written informed consent will be obtained from each parent of the children included in the study stating they accepted the treatment. The study will be performed among children aged 7 to 9 years and who required inferior alveolar block for their treatment. Children who needed anaesthesia for dental treatment will be randomly divided into two groups Group A and Group B using a lottery randomization technique. control group: the children in this group will be delivered Inferior alveolar nerve block in a conventional way [1 min of topical anaesthesia and local infiltration] Experimental group: A Buzzy external cold and vibrating device will be used on the site of application [right/left face] 2 minutes before anaesthesia and this application will be maintained throughout the injection.

At the first visit, the children in Group A will receive the control intervention and those in group B will receive the experimental intervention. A wash out period of 7 days was observed, after which the second visit will be scheduled. At the second visit, the children in Group A will receive the experimental intervention and Group B will receive the control intervention. Demographic details, informed consent from the parents, and assent from the children will be obtained before the commencement of the study. Outcomes will be recorded as primary and secondary outcomes. primary outcomes includes FLACC, WBS and parental scale where as secondary outcomes will be pulse rate and Frankel behaviour rating scale.

Pulse rate will be recorded before anaesthesia, during anaesthesia and 1 min after delivery of anaesthesia, Frankel behaviour rating scale will be measured before, during and after anaesthesia procedures. FLACC and WBS scales will be used to objectively and subjectively record the pain perception. parental scale will be used to determine parental view regarding pain scale during anaesthesia procedure.

ELIGIBILITY:
Inclusion criteria

1. Healthy children with no systemic illness, allergies
2. Co-operative child
3. Patient requiring block for dental treatment
4. children with proper parental consent Exclusion criteria

1. Children with systemic illness and allergy 2. Un co-operative child

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
SEM | During the delivery of anesthesia
  Sound, Eye, Motor
WBS | During the delivery of anesthesia
  WONG BAKER SCALE
parental scale | after administration of anesthesia
  PARENTAL SCALE

SECONDARY OUTCOMES:
PULSE RATE | Measured three times. 15 minutes before the delivery of anesthesia, b. At the time of delivery of anesthesia and c. 1 minute after the delivery of anesthesia
  Pulse rate examined with a pulse oximeter
BEHAVIOURAL RATING SCALE | Measured three times. 15 minutes before the delivery of anesthesia, b. At the time of delivery of anesthesia and c. 1 minute after the delivery of anesthesia
  Behaviour was measured using behaviour rating scale either definitely negative, negative, positive or positive behaviour

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Jizan, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No